CLINICAL TRIAL: NCT03536884
Title: A Multicenter, Randomized, Double-Blind, Secukinumab-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab Compared to an Active Comparator in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Acronym: BE RADIANT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0015; 2017-003784-35 (EudraCT Number)
Record Dates: First submitted 2018-05-14; First posted 2018-05-25 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Chronic Plaque Psoriasis; Moderate to Severe Chronic Plaque Psoriasis
Keywords: Bimekizumab; PSO; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab; secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bimekizumab dosage regimen 1 (Experimental): Subjects randomized to this arm will receive bimekizumab dosage regimen 1 (BKZ 1).
  At Week 16 subjects will be re-randomized and continue to receive BKZ 1 or to switch to bimekizumab regimen 2 (BKZ 2).
  Placebo will be administered at pre-specified time-points to maintain the blinding over the double-blind Treatment Period.
  Subjects allowed to enroll in the open-label extension (OLE) Period will receive BKZ 1 or BKZ 2. Subjects will switch from BKZ 1 to BKZ 2 at Week 64 or at the next scheduled Visit.
  Eligible subjects who completed OLE, have entered Safety Follow Up (SFU) or completed SFU would start OLE2 on BKZ 1 before switching to BKZ 2 after 16 weeks or start OLE2 on BKZ 2.
  Interventions: Drug: Bimekizumab; Other: Placebo
- Bimekizumab dosage regimen 2 (Experimental): Subjects randomized to this arm will receive bimekizumab dosage regimen 2 (BKZ 2) starting at Week 16 after initial treatment on bimekizumab regimen 1 (BKZ 1) for 16 weeks.
  Placebo will be administered at pre-specified time-points to maintain the blinding over the double-blind Treatment Period.
  Subjects allowed to enroll in the open-label extension (OLE) Period will receive BKZ 1 or BKZ 2. Subjects will switch from BKZ 1 to BKZ 2 at Week 64 or at the next scheduled Visit.
  Eligible subjects who completed OLE, have entered SFU or completed SFU would start OLE2 on BKZ 1 before switching to BKZ 2 after 16 weeks or start OLE2 on BKZ 2.
  Interventions: Drug: Bimekizumab; Other: Placebo
- Secukinumab (Active Comparator): Subjects will receive secukinumab. Subjects allowed to enroll in the open-label extension (OLE) Period will be re-randomized to receive bimekizumab dosage regimen 1 (BKZ 1) or bimekizumab dosage regimen 2 (BKZ 2).
  Eligible subjects who completed OLE, have entered SFU or completed SFU would start OLE2 on BKZ 1 before switching to BKZ 2 after 16 weeks or start OLE2 on BKZ 2.
  Interventions: Drug: Bimekizumab; Drug: Secukinumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: UCB4940
Drug: Secukinumab — Subjects will receive secukinumab at pre-specified time-points.
  Other Names: COSENTYX®
  Arms: Secukinumab
Other: Placebo — Subjects will receive placebo at pre-specified time-points to maintain the blinding in the double-blind Treatment Period.
  Other Names: PBO
  Arms: Bimekizumab dosage regimen 1; Bimekizumab dosage regimen 2

SUMMARY:
This is a study to compare the efficacy of bimekizumab versus secukinumab in subjects with moderate to severe chronic plaque psoriasis (PSO).

DETAILED DESCRIPTION:
The study consists of a 48-week double-blind Treatment Period, an optional 96-week open-label extension (OLE) Period and an optional 48-week OLE2 Period for eligible subjects in the USA and Canada.

ELIGIBILITY:
Inclusion Criteria:

Double-blind Treatment Period

* Male or female at least 18 years of age
* Subject must have had chronic plaque psoriasis (PSO) for at least 6 months prior to the Screening visit
* Subject must have Psoriasis Area Severity Index (PASI) >=12 and body surface area (BSA) affected by PSO >=10% and Investigator's Global Assessment (IGA) score >=3 on a 5 point scale
* Subject must be a candidate for systemic PSO therapy and/or phototherapy
* Subject must be considered, in the opinion of the Investigator, to be a suitable candidate for treatment with secukinumab per regional labeling and has no contraindications to receive secukinumab as per the local label
* Female subject of childbearing potential must be willing to use highly effective method of contraception

Open-label extension (OLE) Period

* Completed the double-blind Treatment Period without meeting any withdrawal criteria
* All Week 48 visit assessments completed
* Compliant with ongoing clinical study requirements
* Signed a separate OLE Period Informed Consent Form (ICF)
* Female subject of childbearing potential must be willing to use highly effective method of contraception

OLE2 Period (USA and Canada)

* Completed the OLE Period without meeting any withdrawal criteria
* Compliant with ongoing clinical study requirements
* Female subject of childbearing potential must be willing to use highly effective method of contraception
* Subjects with a diagnosis of Crohn's disease or ulcerative colitis are allowed as long as they have no active symptomatic disease (US only)
* Signed a separate OLE2 Period ICF

Exclusion Criteria:

Double-blind Treatment Period

* Subject has an active infection (except common cold), a serious infection, or a history of opportunistic, recurrent or chronic infections
* Subject has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Subject has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection
* Subject has any other condition, including medical or psychiatric, which, in the Investigator's judgment, would make the subject unsuitable for inclusion in the study
* Presence of active suicidal ideation or severe depression
* Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer

OLE2 Period (USA and Canada)

* Subject has developed any medical or psychiatric condition, which, in the Investigator's judgment, would make the subject unsuitable for inclusion in OLE2 Period
* Subject had a positive or indeterminate interferon-gamma release assay (IGRA) in the OLE study to Week 144, unless appropriately evaluated and treated
* Presence of active suicidal ideation or severe depression
* Subject has developed any active malignancy or history of malignancy prior to the OLE2 Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (77):
- United States (25):
  - Ps0015 975, Santa Ana, California
  - Ps0015 939, Danbury, Connecticut
  - Ps0015 903, Ocala, Florida
  - Ps0015 921, Ormond Beach, Florida
  - Ps0015 977, Pembroke Pines, Florida
  - Ps0015 936, Tampa, Florida
  - Ps0015 976, Tampa, Florida
  - Ps0015 970, West Palm Beach, Florida
  - Ps0015 966, Sandy Springs, Georgia
  - Ps0015 954, Skokie, Illinois
  - Ps0015 972, West Dundee, Illinois
  - Ps0015 900, West Des Moines, Iowa
  - Ps0015 944, New Orleans, Louisiana
  - Ps0015 915, Clayton, Missouri
  - Ps0015 953, St Louis, Missouri
  - Ps0015 901, Portsmouth, New Hampshire
  - Ps0015 965, Kew Gardens, New York
  - Ps0015 969, High Point, North Carolina
  - Ps0015 971, Wilmington, North Carolina
  - Ps0015 980, Bexley, Ohio
  - Ps0015 920, Portland, Oregon
  - Ps0015 929, Portland, Oregon
  - Ps0015 979, Dallas, Texas
  - Ps0015 924, Houston, Texas
  - Ps0015 978, Pflugerville, Texas
- Australia (5):
  - PS0015 3, Carlton
  - PS0015 7, Hectorville
  - PS0015 6, Kogarah
  - Ps0015 11, Parkville
  - PS0015 9, Woolloongabba
- Belgium (3):
  - Ps0015 50, Brussels
  - Ps0015 54, Brussels
  - Ps0015 52, Liège
- Canada (7):
  - Ps0015 673, Halifax
  - Ps0015 671, Hamilton
  - Ps0015 663, Mississauga
  - Ps0015 661, Peterborough
  - Ps0015 678, Richmond Hill
  - Ps0015 677, Toronto
  - Ps0015 657, Waterloo
- Ps0015 153, Toulouse, France
- Germany (11):
  - Ps0015 223, Augsburg
  - Ps0015 237, Berlin
  - Ps0015 211, Hamburg
  - Ps0015 215, Lübeck
  - Ps0015 213, Mahlow
  - Ps0015 238, Mainz
  - Ps0015 234, München
  - Ps0015 219, Münster
  - Ps0015 236, Neu-Ulm
  - Ps0015 222, Tübingen
  - Ps0015 204, Witten
- Netherlands (2):
  - Ps0015 265, Amsterdam
  - Ps0015 263, Breda
- Poland (12):
  - Ps0015 355, Bialystok
  - Ps0015 361, Bialystok
  - Ps0015 369, Bialystok
  - Ps0015 352, Gdansk
  - Ps0015 366, Katowice
  - Ps0015 378, Katowice
  - Ps0015 376, Krakow
  - Ps0015 379, Krakow
  - Ps0015 372, Lodz
  - Ps0015 377, Ostrowiec Świętokrzyski
  - Ps0015 368, Wroclaw
  - Ps0015 375, Wroclaw
- Spain (6):
  - Ps0015 455, Alicante
  - Ps0015 450, Barcelona
  - Ps0015 451, Madrid
  - Ps0015 454, Madrid
  - Ps0015 456, Madrid
  - Ps0015 457, Sant Joan Despí
- Turkey (Türkiye) (3):
  - Ps0015 763, Gaziantep
  - Ps0015 762, Istanbul
  - Ps0015 760, Kayseri
- United Kingdom (2):
  - Ps0015 559, Newcastle upon Tyne
  - Ps0015 555, Salford

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Result] Strober B, Paul C, Blauvelt A, Thaci D, Puig L, Lebwohl M, White K, Vanvoorden V, Deherder D, Gomez NN, Eyerich K. Bimekizumab efficacy and safety in patients with moderate to severe plaque psoriasis: Two-year interim results from the open-label extension of the randomized BE RADIANT phase 3b trial. J Am Acad Dermatol. 2023 Sep;89(3):486-495. doi: 10.1016/j.jaad.2023.04.063. Epub 2023 May 12. PMID 37182701
- [Result] Lebwohl M, Merola JF, Strober B, Armstrong A, Yoshizaki A, Gisondi P, Szilagyi B, Peterson L, de Cuyper D, Cross N, Davies O, Gottlieb AB. Bimekizumab safety in moderate to severe plaque psoriasis: Rates of hepatic events and changes in liver parameters over 2 years in randomized phase 3/3b trials. J Am Acad Dermatol. 2024 Aug;91(2):281-289. doi: 10.1016/j.jaad.2024.03.041. Epub 2024 Apr 6. PMID 38588819
- [Result] Merola JF, Gottlieb AB, Pinter A, Elewski B, Gooderham M, Warren RB, Piaserico S, Wixted K, Cross N, Tilt N, Wiegratz S, Mrowietz U. Bimekizumab Efficacy in High-Impact Areas: Pooled 2-Year Analysis in Scalp, Nail, and Palmoplantar Psoriasis from Phase 3/3b Randomized Controlled Trials. Dermatol Ther (Heidelb). 2024 Dec;14(12):3291-3306. doi: 10.1007/s13555-024-01295-w. Epub 2024 Nov 22. PMID 39578348
- [Result] Strober B, Boehncke WH, Krueger JG, Magnolo N, Vender R, Warren RB, Lopez Pinto JM, Kavanagh S, Hoepken B, Gisondi P. Bimekizumab Efficacy in Psoriasis by Subgroups: Post Hoc Analysis of Phase 3/3b Clinical Trials. Dermatol Ther (Heidelb). 2025 Dec;15(12):3633-3650. doi: 10.1007/s13555-025-01557-1. Epub 2025 Oct 8. PMID 41060492
- [Derived] Merola JF, Warren RB, Thaci D, Gordon KB, Nishida E, Strober B, Conrad C, Kavanagh S, Lopez Pinto JM, Hoepken B, Gisondi P. Bimekizumab Complete Clearance of Both Skin and Nail Psoriasis: Comparative Efficacy in Phase III/IIIb Studies. Am J Clin Dermatol. 2025 Nov;26(6):967-979. doi: 10.1007/s40257-025-00968-2. Epub 2025 Aug 31. PMID 40886218
- [Derived] Warren RB, Lebwohl M, Thaci D, Gooderham M, Pinter A, Paul C, Gisondi P, Szilagyi B, White K, Deherder D, Staelens F, Lambert J, Strober B. Bimekizumab efficacy and safety through 3 years in patients with moderate-to-severe plaque psoriasis: long-term results from the BE RADIANT phase IIIb trial open-label extension period. Br J Dermatol. 2025 Jun 20;193(1):44-55. doi: 10.1093/bjd/ljaf032. PMID 39862230
- [Derived] Augustin M, Gottlieb AB, Lebwohl M, Pinter A, Warren RB, Puig L, Warham R, Lambert J, Wiegratz S, Szilagyi B, Blauvelt A. Complete Skin Clearance is Associated with the Greatest Benefits to Health-Related Quality of Life and Perceived Symptoms for Patients with Psoriasis. Dermatol Ther (Heidelb). 2024 Oct;14(10):2841-2857. doi: 10.1007/s13555-024-01261-6. Epub 2024 Sep 17. PMID 39285121
- [Derived] Kokolakis G, Warren RB, Strober B, Blauvelt A, Puig L, Morita A, Gooderham M, Korber A, Vanvoorden V, Wang M, de Cuyper D, Madden C, Nunez Gomez N, Lebwohl M. Bimekizumab efficacy and safety in patients with moderate-to-severe plaque psoriasis who switched from adalimumab, ustekinumab or secukinumab: results from phase III/IIIb trials. Br J Dermatol. 2023 Feb 22;188(3):330-340. doi: 10.1093/bjd/ljac089. PMID 36751950
- [Derived] Gottlieb AB, Warren RB, Augustin M, Garcia L, Cioffi C, Peterson L, Pelligra C, Ciaravino V. Psychometric Validation of the Psoriasis Symptoms and Impacts Measure (P-SIM): A Novel Patient-Reported Outcome Instrument for Patients with Plaque Psoriasis, Using Reported Data from the BE RADIANT Phase 3b Trial. Adv Ther. 2021 Oct;38(10):5253-5269. doi: 10.1007/s12325-021-01836-1. Epub 2021 Sep 2. PMID 34471992
- [Derived] Yeremenko N. Out of the shadow of interleukin-17A: the role of interleukin-17F and other interleukin-17 family cytokines in spondyloarthritis. Curr Opin Rheumatol. 2021 Jul 1;33(4):333-340. doi: 10.1097/BOR.0000000000000805. PMID 34001692
- [Derived] Reich K, Warren RB, Lebwohl M, Gooderham M, Strober B, Langley RG, Paul C, De Cuyper D, Vanvoorden V, Madden C, Cioffi C, Peterson L, Blauvelt A. Bimekizumab versus Secukinumab in Plaque Psoriasis. N Engl J Med. 2021 Jul 8;385(2):142-152. doi: 10.1056/NEJMoa2102383. Epub 2021 Apr 23. PMID 33891380
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Product Information — https://www.ema.europa.eu/en/documents/product-information/bimzelx-epar-product-information_en.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in June 2018 and concluded in August 2023. Study has Screening Period (2-5 weeks (wk)), DB Treatment Period 48 wks (ITP-Wk 0-16 and MTP- Wk 16-Wk 48), an optional OLE Period (96 wks) followed by SFU Visit (20 wks after final dose) and an optional OLE2 Period followed by SFU2 Visit (20 wks after final dose).
Pre-assignment Details: Participant flow refers to the Randomized Set (RS), Maintenance Set (MS), Open-Label Set (OLS), and Open-Label Set 2 (OLS2).
Groups:
- ITP: Bimekizumab (BKZ) 320 Milligrams (mg) Q4W: Participants randomized to this arm received BKZ 320 mg subcutaneously (sc) every 4 weeks (Q4W) for 16 weeks in the Initial Treatment Period (ITP). Placebo was administered at pre-specified time-points to maintain the blinding.
- ITP: Secukinumab 300 mg Q4W: Participants received secukinumab 300 mg sc at Baseline and Weeks 1, 2, 3, and 4 followed by dosing Q4W until Week 16 in the Initial Treatment Period.
- MTP: BKZ 320 mg Q4W/Q8W: Participants randomized to this arm received BKZ 320 mg sc Q4W for 16 weeks in the Initial Treatment Period. At Week 16, participants were re-randomized to receive BKZ 320 mg sc Q8W until Week 48 in the Maintenance Treatment Period (MTP). Placebo was administered at pre-specified time-points to maintain the blinding.
- MTP: BKZ 320 mg Q4W/Q4W: Participants randomized to this arm received BKZ 320 mg sc Q4W for 16 weeks in the Initial Treatment Period. At Week 16, participants continued to receive BKZ 320 mg sc every 4 Weeks (Q4W/Q4W) until Week 48 in the Maintenance Treatment Period.
- MTP: Secukinumab 300 mg Q4W/Q4W: Participants in secukinumab arm continued to receive secukinumab 300 mg sc Q4W until Week 48 in the Maintenance Treatment Period.
- OLE Period: BKZ Week 0-48/BKZ Q8W 320 mg: Participants randomized to this arm received BKZ 320 mg sc Q4W for the first 16 weeks and then re-randomized to receive BKZ 320 mg sc Q4W or Q8W until Week 48 of the double-blind Treatment Period. Based on the PASI90 response and the dose the participant was receiving at Week 48, participants were randomized to receive BKZ 320 mg sc Q8W until Week 136 in the Open-Label Extension (OLE) Period.
- OLE Period: BKZ Week 0-48/ BKZ Q4W 320 mg: Participants randomized to this arm received BKZ 320 mg sc Q4W for the first 16 weeks and then re-randomized to receive BKZ 320 mg sc Q4W or Q8W until Week 48 of the double-blind Treatment Period. Based on the PASI90 response and the dose the participant was receiving at Week 48, participants were randomized to receive BKZ 320 mg sc Q4W starting in OLE Period. The participant's dosing interval was changed from BKZ 320mg Q4W to BKZ 320mg Q8W at Week 64, or at the next scheduled clinic visit if the participant has already completed the Week 64 after protocol amendment 5.
- OLE Period: Secukinumab Week 0-48/ BKZ Q8W 320 mg: Participants randomized to this arm received Secukinumab 300 mg sc Q4W until Week 48 of the double-blind Treatment Period. Based on the PASI90 response in double-blind Treatment Period, participants randomized to receive BKZ 320 mg sc Q8W until Week 136 of the OLE Period.
- OLE Period: Secukinumab Week 0-48/ BKZ Q4W 320 mg: Participants randomized to this arm received Secukinumab 300 mg sc Q4W until Week 48 of the double-blind Treatment Period. Based on the PASI90 response in double-blind Treatment Period, participants randomized to receive BKZ 320 mg sc Q4W starting in OLE Period. The participant's dosing interval was changed from BKZ 320mg Q4W to BKZ 320mg Q8W at Week 64, or at the next scheduled clinic visit if the participant has already completed the Week 64 after protocol amendment 5.
- OLE2 Period - Group A: BKZ 320 mg Q8W: Participants who were still receiving treatment in the OLE Period and attended the Week 144 visit were directly rolled over to the OLE2 Period. In OLE2 Period, participants continued receiving BKZ 320 mg sc Q8W for 40 additional weeks until OLE2 Week 48.
- OLE2 Period - Group B: BKZ 320 mg Q8W: Participants who completed the Week 144 and were participating in the Safety Follow-Up (SFU) or had completed the SFU visit reinitiated their treatment in the OLE2 Period after having undergone Screening assessments during a 4-week OLE2 Screening Period. Participants with an IGA score less than (<) 3 at the Week 144/OLE2 Baseline Visit continued receiving BKZ 320 mg sc Q8W for 40 additional weeks until OLE2 Week 48 in OLE2 Period.
- OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W: Participants who completed the Week 144 visit and were participating in the SFU or had completed the SFU visit reinitiated their treatment in the OLE2 Period after having undergone Screening assessments during a 4-week OLE2 Screening Period. Participants with an IGA score greater than or equal to (>=) 3 at the Week 144/OLE2 Baseline Visit received BKZ 320 mg sc Q4W for the first 16 weeks, and then switched to BKZ 320 mg sc Q8W for 24 weeks until OLE2 Week 48 in OLE2 Period.
Period: Double-Blind (DB) Period: ITP Wk 0-16
Arm/Group | ITP: Bimekizumab (BKZ) 320 Milligrams (mg) Q4W | ITP: Secukinumab 300 mg Q4W | MTP: BKZ 320 mg Q4W/Q8W | MTP: BKZ 320 mg Q4W/Q4W | MTP: Secukinumab 300 mg Q4W/Q4W | OLE Period: BKZ Week 0-48/BKZ Q8W 320 mg | OLE Period: BKZ Week 0-48/ BKZ Q4W 320 mg | OLE Period: Secukinumab Week 0-48/ BKZ Q8W 320 mg | OLE Period: Secukinumab Week 0-48/ BKZ Q4W 320 mg | OLE2 Period - Group A: BKZ 320 mg Q8W | OLE2 Period - Group B: BKZ 320 mg Q8W | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W
Started | 373 | 370 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 362 | 354 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 8 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unblinding was reason for dropout | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawn by Investigator for abnormal lab values | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unable to attend visits | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-Blind Period: MTP Wk 16-48
Arm/Group | ITP: Bimekizumab (BKZ) 320 Milligrams (mg) Q4W | ITP: Secukinumab 300 mg Q4W | MTP: BKZ 320 mg Q4W/Q8W | MTP: BKZ 320 mg Q4W/Q4W | MTP: Secukinumab 300 mg Q4W/Q4W | OLE Period: BKZ Week 0-48/BKZ Q8W 320 mg | OLE Period: BKZ Week 0-48/ BKZ Q4W 320 mg | OLE Period: Secukinumab Week 0-48/ BKZ Q8W 320 mg | OLE Period: Secukinumab Week 0-48/ BKZ Q4W 320 mg | OLE2 Period - Group A: BKZ 320 mg Q8W | OLE2 Period - Group B: BKZ 320 mg Q8W | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W
Started | 0 | 0 | 215 | 147 | 354 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 205 | 138 | 325 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 10 | 9 | 29 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 3 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: OLE Period: Wk48-Wk144
Arm/Group | ITP: Bimekizumab (BKZ) 320 Milligrams (mg) Q4W | ITP: Secukinumab 300 mg Q4W | MTP: BKZ 320 mg Q4W/Q8W | MTP: BKZ 320 mg Q4W/Q4W | MTP: Secukinumab 300 mg Q4W/Q4W | OLE Period: BKZ Week 0-48/BKZ Q8W 320 mg | OLE Period: BKZ Week 0-48/ BKZ Q4W 320 mg | OLE Period: Secukinumab Week 0-48/ BKZ Q8W 320 mg | OLE Period: Secukinumab Week 0-48/ BKZ Q4W 320 mg | OLE2 Period - Group A: BKZ 320 mg Q8W | OLE2 Period - Group B: BKZ 320 mg Q8W | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W
Started | 0 | 0 | 0 | 0 | 0 | 238 (Participants who provided consent to continue in OLE Period.) | 98 (Participants who provided consent to continue in OLE Period.) | 122 (Participants who provided consent to continue in OLE Period.) | 196 (Participants who provided consent to continue in OLE Period.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 205 | 80 | 106 | 167 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 33 | 18 | 16 | 29 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 10 | 8 | 6 | 13 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 1 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 12 | 7 | 6 | 6 | 0 | 0 | 0
Not completed — Not dosing for over 6 Months while out of country | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient held IP due to pandemic, not restarted | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Went to jail, unable to continue study visits | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — She wants to be pregnant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: OLE2 Period: Wk 144/OLE2 BL- OLE2 Wk 48
Arm/Group | ITP: Bimekizumab (BKZ) 320 Milligrams (mg) Q4W | ITP: Secukinumab 300 mg Q4W | MTP: BKZ 320 mg Q4W/Q8W | MTP: BKZ 320 mg Q4W/Q4W | MTP: Secukinumab 300 mg Q4W/Q4W | OLE Period: BKZ Week 0-48/BKZ Q8W 320 mg | OLE Period: BKZ Week 0-48/ BKZ Q4W 320 mg | OLE Period: Secukinumab Week 0-48/ BKZ Q8W 320 mg | OLE Period: Secukinumab Week 0-48/ BKZ Q4W 320 mg | OLE2 Period - Group A: BKZ 320 mg Q8W | OLE2 Period - Group B: BKZ 320 mg Q8W | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 (Participants who provided consent to continue in OLE2 Period.) | 66 (Participants who provided consent to continue in OLE2 Period.) | 59 (Participants who provided consent to continue in OLE2 Period.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 61 | 52
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Not completed — Site's business is closing on 30 September 2022 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Site closure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Subject had threatening behavior to site staff | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS) which consisted of all randomized study participants.
Arm/Group | ITP: Bimekizumab (BKZ) 320 Milligrams (mg) Q4W | ITP: Secukinumab 300 mg Q4W | Total Title
Number analyzed (Participants) | 373 | 370 | 743
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 7 | 10
  Between 18 and 65 years | 332 | 324 | 656
  >=65 years | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (14.2) | 44.0 (14.7) | 45.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 135 | 257
  Male | 251 | 235 | 486
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 10 | 9 | 19
  Black | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 347 | 348 | 695
  Other or Mixed | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 32 | 51
  Not Hispanic or Latino | 354 | 338 | 692

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 100 (PASI100) Response at Week 16
Description: The PASI100 response assessments are based on 100% improvement in PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Groups:
- ITP: Bimekizumab (BKZ) 320 mg Q4W: Participants randomized to this arm received BKZ 320 mg sc Q4W for 16 weeks in the Initial Treatment Period (ITP). Placebo was administered at pre-specified time-points to maintain the blinding.
Arm/Group | ITP: Bimekizumab (BKZ) 320 mg Q4W | ITP: Secukinumab 300 mg Q4W
Number analyzed (Participants) | 373 | 370
percentage of participants | 61.7 | 48.9
Statistical Analysis 1: Comparison: ITP: Bimekizumab (BKZ) 320 mg Q4W vs ITP: Secukinumab 300 mg Q4W; Risk Difference: BKZ-Secukinumab calculated using stratified Cochran-Mantel-Haenszel (CMH); Test type: Non-Inferiority — The evaluation of noninferiority is tested at a 1-sided alpha level of 0.025 and based on a 1-sided 97.5% CI and a noninferiority margin of 10%; Risk Difference (RD) = 12.682, 95% CI 2-sided [5.771 to 19.592]
Statistical Analysis 2: Comparison: ITP: Bimekizumab (BKZ) 320 mg Q4W vs ITP: Secukinumab 300 mg Q4W; Odds ratio calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups are based on the CMH test for the general association; Odds Ratio (OR) = 1.714, 95% CI 2-sided [1.271 to 2.310]

2. Secondary Outcome: Percentage of Participants With a PASI75 Response at Week 4
Description: The PASI75 response assessments are based on at least 75% improvement in PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of body areas and converting to 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 4
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | ITP: Bimekizumab (BKZ) 320 mg Q4W | ITP: Secukinumab 300 mg Q4W
Number analyzed (Participants) | 373 | 370
percentage of participants | 71.0 | 47.3
Statistical Analysis 1: Comparison: ITP: Bimekizumab (BKZ) 320 mg Q4W vs ITP: Secukinumab 300 mg Q4W; Odds ratio calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups are based on the CMH test from the general association. P-values are not controlled for multiplicity and should only be considered descriptively; Odds Ratio (OR) = 2.817, 95% CI 2-sided [2.068 to 3.836]

3. Secondary Outcome: Percentage of Participants With a PASI90 Response at Week 16
Description: The PASI90 response assessments are based on at least 90% improvement in PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI=average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | ITP: Bimekizumab (BKZ) 320 mg Q4W | ITP: Secukinumab 300 mg Q4W
Number analyzed (Participants) | 373 | 370
percentage of participants | 85.5 | 74.3

4. Secondary Outcome: Percentage of Participants With a PASI100 Response at Week 48
Description: as for outcome 1
Time Frame: Week 48
Population: The Randomized Set (RS) consisted of all randomized study participants. The Maintenance Set (MS) consisted of all study participants that received at least 1 dose of IMP at Week 16 or later in the Double-Blind Treatment Period (including the Week 16 dose).
Measure: Number; unit: percentage of participants
Groups:
- ITP+MTP: BKZ Q4W/Q4W +BKZ Q4W/Q8W: Participants randomized to this arm received BKZ 320 mg sc Q4W for 16 weeks in the ITP. At Week 16, participants either continued to receive BKZ 320 mg sc every 4 Weeks (Q4W/Q4W) or re-randomized to receive BKZ 320 mg sc Q8W until Week 48 in the MTP. Placebo was administered at pre-specified time-points to maintain the blinding.
- ITP+MTP: Secukinumab 300 mg Q4W/Q4W: Participants received secukinumab 300 mg sc at Baseline and Weeks 1, 2, 3, and 4 followed by dosing Q4W until Week 16 in the ITP. Participants continued to receive secukinumab 300 mg sc Q4W until Week 48 in the MTP.
Arm/Group | ITP+MTP: BKZ Q4W/Q4W +BKZ Q4W/Q8W | ITP+MTP: Secukinumab 300 mg Q4W/Q4W | MTP: BKZ 320 mg Q4W/Q8W | MTP: BKZ 320 mg Q4W/Q4W | MTP: Secukinumab 300 mg Q4W/Q4W
Number analyzed (Participants) | 373 | 370 | 215 | 147 | 354
percentage of participants | 67.3 | 46.2 | 66.5 | 73.5 | 48.3
Statistical Analysis 1: Comparison: ITP+MTP: BKZ Q4W/Q4W +BKZ Q4W/Q8W vs ITP+MTP: Secukinumab 300 mg Q4W/Q4W; Odds ratio calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.490, 95% CI 2-sided [1.835 to 3.377]
Statistical Analysis 2: Comparison: MTP: BKZ 320 mg Q4W/Q8W vs MTP: Secukinumab 300 mg Q4W/Q4W; Odds ratio calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups are based on the CMH test from the general association; Odds Ratio (OR) = 2.168, 95% CI 2-sided [1.511 to 3.110]
Statistical Analysis 3: Comparison: MTP: BKZ 320 mg Q4W/Q4W vs MTP: Secukinumab 300 mg Q4W/Q4W; Odds ratio calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups are based on the CMH test from the general association; Odds Ratio (OR) = 3.243, 95% CI 2-sided [2.103 to 5.000]

5. Secondary Outcome: Percentage of Participants With a Investigator´s Global Assessment (IGA) Response (0/1) at Week 16
Description: The IGA measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as Clear (0) or Almost Clear (1) with at least a two-category improvement from Baseline at Week 16.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | ITP: Bimekizumab (BKZ) 320 mg Q4W | ITP: Secukinumab 300 mg Q4W
Number analyzed (Participants) | 373 | 370
percentage of participants | 85.5 | 78.6

6. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Adjusted by Duration of Participant Exposure to Investigational Medicinal Product (IMP) From Baseline up to Week 225
Description: The number of TEAEs adjusted by duration of exposure to study treatment was scaled such that provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline up to Week 225
Population: The Safety Set (SS) consisted of all study participants that received at least 1 dose of IMP. The Open-Label Set (OLS) consisted of all study participants who received at least 1 dose of BKZ at Week 48 or later in the OLE Period (including the Week 48 dose). The Open-Label Set 2 (OLS2) consisted of all study participants who received at least 1 dose of BKZ at the Week 144/OLE2 Baseline Visit or later in the OLE2 Period (including the Week 144/OLE2 Baseline dose).
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- MTP: BKZ 320 mg Q8W (Week 16 to Week 48): Participants who received at least one dose of BKZ 320 mg sc Q8W from Week 16 until Week 48.
- ITP+MTP: BKZ 320 mg Q4W (up to Week 48): Participants who received at least one dose of BKZ 320 mg sc Q4W until Week 48.
- ITP+MTP: Secukinumab 300 mg Q4W (up to Week 48): Participants received secukinumab 300 mg sc at Baseline and Weeks 1, 2, 3, and 4 followed by dosing Q4W until Week 48.
- OLE Period: BKZ 320 mg Q8W (Week 48 to Week 144): Participants received BKZ 320 mg sc Q8W from Week 48 until Week 136 during OLE Period. For participants that received both BKZ 320 mg Q4W and Q8W, events are counted in the dose group most recently received prior to the date of the event or assessment.
- OLE Period: BKZ 320 mg Q4W (Week 48 to Week 144): Participants received BKZ 320 mg sc Q4W from Week 48 until Week 136 during OLE Period. The participant's dosing interval was changed from BKZ 320 mg Q4W to BKZ 320 mg Q8W at Week 64, or at the next scheduled clinic visit if the participant has already completed the Week 64.
Arm/Group | MTP: BKZ 320 mg Q8W (Week 16 to Week 48) | ITP+MTP: BKZ 320 mg Q4W (up to Week 48) | ITP+MTP: Secukinumab 300 mg Q4W (up to Week 48) | OLE Period: BKZ 320 mg Q8W (Week 48 to Week 144) | OLE Period: BKZ 320 mg Q4W (Week 48 to Week 144) | OLE2 Period - Group A: BKZ 320 mg Q8W | OLE2 Period - Group B: BKZ 320 mg Q8W | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W
Number analyzed (Participants) | 215 | 373 | 370 | 626 | 294 | 9 | 66 | 59
no. of new events per 100 subject-years | 250.13 [213.09 to 291.75] | 331.26 [293.40 to 372.66] | 234.88 [209.22 to 262.83] | 115.35 [105.27 to 126.14] | 165.22 [143.73 to 189.02] | 164.95 [66.32 to 339.86] | 74.25 [51.72 to 103.26] | 94.18 [65.97 to 130.39]

7. Secondary Outcome: Number of Serious Adverse Events (SAEs) Adjusted by Duration of Participant Exposure to IMP From Baseline up to Week 225
Description: The number of SAEs adjusted by duration of exposure to study treatment was scaled such that it provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline up to Week 225
Population: The SS consisted of all study participants that received at least 1 dose of IMP. The OLS consisted of all study participants who received at least 1 dose of BKZ at Week 48 or later in the OLE Period (including the Week 48 dose). The OLS2 consisted of all study participants who received at least 1 dose of BKZ at the Week 144/OLE2 Baseline Visit or later in the OLE2 Period (including the Week 144/OLE2 Baseline dose).
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- OLE Period: BKZ 320 mg Q8W (Week 48 to Week 144): Participants received BKZ 320 mg sc Q8W from Week 48 until Week 136 during OLE Period. For subjects that received both BKZ 320mg Q4W and Q8W, events are counted in the dose group most recently received prior to the date of the event or assessment.
Arm/Group | MTP: BKZ 320 mg Q8W (Week 16 to Week 48) | ITP+MTP: BKZ 320 mg Q4W (up to Week 48) | ITP+MTP: Secukinumab 300 mg Q4W (up to Week 48) | OLE Period: BKZ 320 mg Q8W (Week 48 to Week 144) | OLE Period: BKZ 320 mg Q4W (Week 48 to Week 144) | OLE2 Period - Group A: BKZ 320 mg Q8W | OLE2 Period - Group B: BKZ 320 mg Q8W | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W
Number analyzed (Participants) | 215 | 373 | 370 | 626 | 294 | 9 | 66 | 59
no. of new events per 100 subject-years | 6.94 [3.17 to 13.17] | 7.33 [4.10 to 12.09] | 6.75 [4.23 to 10.22] | 5.93 [4.48 to 7.70] | 4.34 [2.16 to 7.76] | 12.28 [0.31 to 68.43] | 1.38 [0.03 to 7.66] | 6.39 [1.74 to 16.37]

8. Secondary Outcome: Number of TEAEs Leading to Withdrawal Adjusted by Duration of Participant Exposure to IMP From Baseline up to Week 225
Description: The number of TEAEs leading to discontinuation adjusted by duration of exposure to study treatment was scaled such that it provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline up to Week 225
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | MTP: BKZ 320 mg Q8W (Week 16 to Week 48) | ITP+MTP: BKZ 320 mg Q4W (up to Week 48) | ITP+MTP: Secukinumab 300 mg Q4W (up to Week 48) | OLE Period: BKZ 320 mg Q8W (Week 48 to Week 144) | OLE Period: BKZ 320 mg Q4W (Week 48 to Week 144) | OLE2 Period - Group A: BKZ 320 mg Q8W | OLE2 Period - Group B: BKZ 320 mg Q8W | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W
Number analyzed (Participants) | 215 | 373 | 370 | 626 | 294 | 9 | 66 | 59
no. of new events per 100 subject-years | 1.51 [0.18 to 5.45] | 5.85 [3.02 to 10.22] | 3.33 [1.66 to 5.96] | 2.56 [1.65 to 3.77] | 3.52 [1.61 to 6.69] | 11.33 [0.29 to 63.10] | 2.76 [0.33 to 9.99] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: From Baseline up to 165 weeks for each study participant not entering the OLE2 Period and up to 225 weeks for participants entering OLE2 Period
Description: TEAEs were defined as those AEs that have a start date on or following the first dose of study treatment through final dose of study treatment + 140 days (covering 20-week SFU period). For participants that switched from BKZ 320 mg Q4W to Q8W, events prior to switch are counted in Q4W group and events after switch are counted in Q8W group.
Groups:
- ITP: BKZ 320 mg Q4W (up to Week 16): Participants randomized to this arm received BKZ 320 mg sc Q4W for 16 weeks in the Initial Treatment Period. Placebo was administered at pre-specified time-points to maintain the blinding.
- ITP: Secukinumab 300 mg Q4W (up to Week 16): Participants received secukinumab 300 mg sc at Baseline and Weeks 1, 2, 3, and 4 followed by dosing Q4W until Week 16 in the Initial Treatment Period.
- OLE2 Period - Group A: BKZ 320 mg Q8W: Participants who were still receiving treatment in the OLE Period and attended the Week 144 visit were directly rolled over to the OLE2 Period. In OLE2 Period, participants continued receiving BKZ 320 mg sc Q8W for 40 additional weeks until OLE2 Week 48. Due to small number of participants, each event met the 5% threshold frequency criteria.
Arm/Group | ITP: BKZ 320 mg Q4W (up to Week 16) | ITP: Secukinumab 300 mg Q4W (up to Week 16) | MTP: BKZ 320 mg Q8W (Week 16 to Week 48) | ITP+MTP: BKZ 320 mg Q4W (up to Week 48) | ITP+MTP: Secukinumab 300 mg Q4W (up to Week 48) | OLE Period: BKZ 320 mg Q8W (Week 48 to Week 144) | OLE Period: BKZ 320 mg Q4W (Week 48 to Week 144) | OLE2 Period - Group A: BKZ 320 mg Q8W | OLE2 Period - Group B: BKZ 320 mg Q8W | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W
All-Cause Mortality (participants affected / at risk) | 0/373 | 0/370 | 1/215 | 0/373 | 2/370 | 3/626 | 1/294 | 0/9 | 0/66 | 1/59
Serious Adverse Events (participants affected / at risk) | 10/373 | 6/370 | 9/215 | 15/373 | 22/370 | 56/626 | 11/294 | 1/9 | 1/66 | 4/59
Other Adverse Events (participants affected / at risk) | 107/373 | 88/370 | 87/215 | 140/373 | 166/370 | 233/626 | 103/294 | 7/9 | 18/66 | 19/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITP: BKZ 320 mg Q4W (up to Week 16) (N=373) | ITP: Secukinumab 300 mg Q4W (up to Week 16) (N=370) | MTP: BKZ 320 mg Q8W (Week 16 to Week 48) (N=215) | ITP+MTP: BKZ 320 mg Q4W (up to Week 48) (N=373) | ITP+MTP: Secukinumab 300 mg Q4W (up to Week 48) (N=370) | OLE Period: BKZ 320 mg Q8W (Week 48 to Week 144) (N=626) | OLE Period: BKZ 320 mg Q4W (Week 48 to Week 144) (N=294) | OLE2 Period - Group A: BKZ 320 mg Q8W (N=9) | OLE2 Period - Group B: BKZ 320 mg Q8W (N=66) | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W (N=59)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otosclerosis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease nodular sclerosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboangiitis obliterans (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITP: BKZ 320 mg Q4W (up to Week 16) (N=373) | ITP: Secukinumab 300 mg Q4W (up to Week 16) (N=370) | MTP: BKZ 320 mg Q8W (Week 16 to Week 48) (N=215) | ITP+MTP: BKZ 320 mg Q4W (up to Week 48) (N=373) | ITP+MTP: Secukinumab 300 mg Q4W (up to Week 48) (N=370) | OLE Period: BKZ 320 mg Q8W (Week 48 to Week 144) (N=626) | OLE Period: BKZ 320 mg Q4W (Week 48 to Week 144) (N=294) | OLE2 Period - Group A: BKZ 320 mg Q8W (N=9) | OLE2 Period - Group B: BKZ 320 mg Q8W (N=66) | OLE2 Period -Group B: BKZ 320 mg Q4W/Q8W (N=59)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 49 (50) | 9 (9) | 2 (2) | 7 (7) | 10 (10)
Nasopharyngitis (Infections and infestations) | 47 (54) | 54 (61) | 33 (40) | 62 (76) | 102 (141) | 62 (85) | 34 (41) | 0 (0) | 3 (3) | 1 (1)
Oral candidiasis (Infections and infestations) | 39 (41) | 4 (4) | 36 (47) | 50 (64) | 11 (16) | 53 (68) | 39 (51) | 0 (0) | 4 (4) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 17 (17) | 21 (25) | 23 (26) | 36 (39) | 35 (46) | 13 (13) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (7) | 7 (8) | 10 (14) | 15 (19) | 22 (30) | 30 (40) | 19 (25) | 1 (1) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 5 (5) | 1 (1) | 1 (1) | 7 (8) | 3 (3) | 11 (12) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Psychiatric evaluation abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (5) | 1 (1) | 3 (3) | 2 (12) | 3 (4) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 3 (4) | 8 (9) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3) | 1 (1) | 5 (6) | 16 (17) | 38 (40) | 5 (7) | 0 (0) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT03536884/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT03536884/SAP_001.pdf